CLINICAL TRIAL: NCT03096327
Title: TEAM (Trial on Efficacy and Quality of Life Among Asthmatic Patient With Montelukast)
Acronym: TEAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PharmEvo Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PE/PK/TEAM/IIT/2017-01
Record Dates: First submitted 2017-03-17; First posted 2017-03-30 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: Quality of Life; Asthma control test; Montelukast; Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Endpoint Classification: Safety/Efficacy Study Intervention Model: Two arm Parallel Assignment Masking: Double Blind Primary Purpose: Prevention
Who Masked: Participant, Care Provider
Masking Description: To ensure double-blind allocation, the sponsor, who is not directly involved in clinical team will use a random number sequence generated by a computer software to allocate the participant to either the treatment or placebo group. Patients who will be randomized to the treatment group will receive 10 mg montelukast. Patients in placebo group will receive identical looking drug (placebo) produced by same manufactured.
  Both products will be packaged in identical plastic bottles identifiable only by the patient allocation number. Patient will be asked to take one montelukast each day. Acceptable compliance will be defined as at least taking medication at least 21 days. The patients will be instructed to leave the remaining tablets in bottle so that they would be counted later.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Montelukast) (Experimental): Aireez contains Montelukast which is a potent and selective blocker of the CysLT1 receptor. For treatment of chronic asthma, montelukast is administered once daily to adults as a 10-mg film-coated tablet, to children aged 6-14 years as a 5-mg chewable tablet, and to children aged 2-5 years as a 4-mg chewable tablet form.
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): Patients in placebo group will receive identical looking drug (placebo) produced by same manufactured.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — Montelukast sodium is a selective blocker of the CysLT1 receptor. For treatment of chronic asthma, montelukast is administered once daily to adults as a 10-mg film-coated tablet, to children aged 6-14 years as a 5-mg chewable tablet, and to children aged 2-5 years as a 4-mg chewable tablet form.
  Other Names: TEAM
  Arms: Intervention (Montelukast)
Drug: Placebo — Patients in placebo group will receive identical looking drug (placebo) produced by same manufactured
  Other Names: TEAM
  Arms: Placebo

SUMMARY:
• To compare the quality of Life using AQLQ (s) questionnaire after 4 weeks of Montelukast.

DETAILED DESCRIPTION:
1.1 Background

Asthma is characterized by airway and lung tissue inflammation and airway hyperresponsiveness (AHR) that leads to recurrent symptoms of wheezing, breathlessness, chest tightness, and coughing. AHR indicates an exaggerated response of the airway to nonspecific stimuli, which results in a temporary airflow limitation, leading to airway obstruction. It remains unknown which factors within the airway of an individual trigger reversible airway obstruction and airway narrowing. The airway epithelium is composed of many interacting structural components and inflammatory cells. The number, activation, and secretory component of inflammatory cells in the airway are altered in the disease. In asthma, the number of eosinophils and T lymphocytes is increased in the subepithelial layer.

The impact of asthma has traditionally been measured in terms of the prevalence of the disease, mortality rates, and levels of healthcare utilisation, particularly hospital admissions. However, the impact of asthma extends beyond these outcomes to include effects on lifestyle, wellbeing, and perceived health status. Adults of working age with asthma have poorer health status and quality of life outcomes than those with no asthma. This effect is independent of confounding by sociodemographic and life style factors and is evident across a range of dimensions of quality of life. In comparison with two other chronic health conditions, asthma has a larger adverse impact on health status and quality of life than diabetes.

1.2. Investigational Agent

Montelukast reversibly inhibits cysteinyl leukotrienes (CysLTs), specifically leukotrienes D4 (LTD4 [3]. LTD4 is the most potent bronchoconstricting agent on a molar basis, but Cys-LTs also have chemoattractive properties for many inflammatory cells (mainly eosinophils), effects on vascular permeability, mucous secretions and sensory nerve activation, and are responsible for part of the pathophysiology of asthma.

1.3. Dose Rational/Risk & Benefit

Montelukast is a potent and selective blocker of the CysLT1 receptor. For treatment of chronic asthma, montelukast is administered once daily to adults as a 10-mg film-coated tablet, to children aged 6-14 years as a 5-mg chewable tablet, and to children aged 2-5 years as a 4-mg chewable tablet form. Given their efficacy, antiinflammatory activity, oral administration, and safety, leukotriene modifiers will play an important role in the treatment of asthmatic patient. Side effects most commonly reported above placebo included headache, otitis media, upper respiratory infection, and pharyngitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Asthma
* Signed Informed Consent

Exclusion Criteria:

* Previous adverse reaction to montelukast or other leukotriene inhibitor;
* History of hyper-eosinophilic disorder other than atopic disease;
* Treatment with montelukast within 4 weeks from randomization;
* Asthma exacerbation or treatment with prednisone/other systemic steroid within 4 weeks from randomization.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
To assess the change in quality of Life using AQLQ (s) questionnaire after 4 weeks of Montelukast. | 0 days to 4 weeks
  [Designated as safety issue: No]

SECONDARY OUTCOMES:
To assess the change in Control of Asthma using AQLQ (s) questionnaire after 4 weeks of Montelukast. | 0 days to 4 weeks
  [Designated as safety issue: No]
Proportion of participants experiencing an adverse event (AE) | 0 days to 4 weeks
  [Designated as safety issue: Yes]

CONTACTS AND LOCATIONS:
Overall Officials: Masood Jawaid, MRCS,FCPS, Study Director — PharmEvo Pvt Ltd
Locations (1):
- Dr. Nadeem Rizvi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No